CLINICAL TRIAL: NCT06668012
Title: A Multicenter, Open, Comparative Study on the Effect of Palomacare® Vaginal Gel on Vaginal Dysbiosis in Premenopausal Women (DISPALOMA)
Brief Title: A Multicenter, Open, Comparative Study on Vaginal Dysbiosis in Premenopausal Women (DISPALOMA)
Acronym: DISPALOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISPALOMA
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Dysbiosis
Keywords: Vaginal; Palomacare; Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: Multicenter, open, comparative study, where all eligible patients with vaginal dysbiosis (vaginal pH >4.5) will be assigned to one of the 3 study groups (1:1:1) according to the randomization list for random assignment to groups B and C:
  A. Symptomatic patients: Treatment with Palomacare® vaginal gel for 6 days B. Asymptomatic patients: Treatment with Palomacare® vaginal gel for 6 days C. Asymptomatic patients: Monitored follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A - Symptomatic patients (Active Comparator): Treatment with Palomacare® vaginal gel for 6 days
  Interventions: Device: Palomacare® vaginal gel is a medical device with CE class IIa.
- B - Asymptomatic patients (Active Comparator): Treatment with Palomacare® vaginal gel for 6 days
  Interventions: Device: Palomacare® vaginal gel is a medical device with CE class IIa.
- C - Asymptomatic patients (No Intervention): Monitored follow-up

INTERVENTIONS:
Device: Palomacare® vaginal gel is a medical device with CE class IIa. — The duration of the study for each patient will be approximately 11-12 days and the treatment for groups A and B will be 6 days.
  In a first pilot study in asymptomatic women, a tendency towards a positive effect on the composition of vaginal fluid was already observed, as assessed by diagnostic tests and classified using a Likert scale. A subsequent study showed that treatment with a different vaginal gel but with an identical concentration of ingredients from Palomacare® vaginal gel, for 21 consecutive days, is able to improve the composition of vaginal fluid.
  Based on these preliminary data, it is possible to hypothesize that the action of Palomacare® vaginal gel will have a positive effect on the composition of vaginal fluid in patients affected by dysbiosis, whether asymptomatic or not.
  Arms: A - Symptomatic patients; B - Asymptomatic patients

SUMMARY:
The hypothesis is raised of improving the status of vagnal microbiota with a non-hormonal topical product in early situations of dysbiosis in which the vaginal pH is elevated and the patient may or may not be symptomatic, in order to try to prevent the appearance of future established vaginal infections.

DETAILED DESCRIPTION:
Multicenter, open, comparative study, where all eligible patients with vaginal dysbiosis (vaginal pH >4.5) will be assigned to one of the 3 study groups (1:1:1) according to the randomization list for random assignment to groups B and C:

A. Symptomatic patients: Treatment with Palomacare® vaginal gel for 6 days B. Asymptomatic patients: Treatment with Palomacare® vaginal gel for 6 days C. Asymptomatic patients: Monitored follow-up

2 visits will be made throughout the study: visit 1 (initial visit, between days 9 and 15 of the menstrual cycle) and visit 2 (final visit, within 5 days after the end of treatment or equivalent in the case of the monitored follow-up group, always before the next menstruation).

The study will consist of two phases; the first phase or PILOT, where 30 patients (10 per group) will be included with the intervention of 2 centers, and a second phase or EXTENSION, where 60 additional patients (20 per group) will be included, obtaining a total of 90 patients (30 per group) at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 45 years of age, inclusive.
2. Who are attending a gynecological visit for any reason and who are in the first phase of the menstrual cycle, between the end of menstruation and before ovulation (approximately between days 9 and 15).
3. With regular menstrual cycles of between 24 and 35 days.
4. Who are able to understand and sign the informed consent after the nature of the study has been fully explained to them.
5. With a vaginal pH higher than 4.5 with or without symptoms

Exclusion Criteria:

1. Diagnosis of another vaginal or vulvar condition that may confuse the interpretation of the response to the investigational product (erosive lichen planus, inflammatory desquamative vaginitis, or contact dermatitis involving the vulvar epithelium).
2. Diagnosis of cervical intraepithelial neoplasia (CIN), cervical carcinoma, or endometrial neoplasia.
3. Active genitourinary infections (VVC, N. gonorrhoeae, C. trachomatis, or T. vaginalis) at the time of inclusion or within 15 days prior to inclusion in the study.
4. Active genital lesions (ulcers or vesicles compatible with herpes or warts) or genital bleeding.
5. Pregnant patients or in the immediate postpartum period (up to 40 days).
6. Contraception with copper IUD.
7. Use of oral or topical antibiotics, or vaginal antifungals in the two weeks prior to the initial visit.
8. Planned immunosuppressive therapy.
9. Decompensated chronic diseases (diabetes, epilepsy, high blood pressure, etc.).
10. Use of any other experimental drug or device during the 30 days prior to selection.
11. Formal contraindication for the use of the product, such as hypersensitivity to any of the components of the study treatments.
12. Inability, at the discretion of the researcher, to comply with the requirements of the study, either due to follow-up problems or due to psychophysical characteristics.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Palomacare® vaginal gel on vaginal microbiota (VM) | Through study completion, an average of 12 days
  To evaluate the effect of Palomacare® vaginal gel on VM, the change in microbial diversity, vaginotype and taxonomic profile of the vaginal microbiome will be analyzed between V1 and V2 in each group.

SECONDARY OUTCOMES:
Effect of Palomacare® vaginal gel on symptoms and pH | Through study completion, an average of 12 days
  To assess the effect of Palomacare® vaginal gel on:
  * Symptoms (amine odour, leucorrhoea and itching): for each symptom an VAS intensity scale will be used and the time to show changes in each of the symptoms will be assessed by directly asking the patient.
  * Vaginal pH: vaginal pH refers to the degree of acidity of the vaginal environment. Adequate vaginal pH levels should be between 3.8 - 4.4. However, these vary throughout the woman's cycle and at different stages of life. The researcher will carry out this measurement at visit 1 and visit 2, noting the numerical value of the patient's vaginal pH.
Satisfaction with the use of Palomacare® vaginal gel | Through study completion, an average of 12 days
  To assess the degree of satisfaction regarding the use of Palomacare® vaginal gel using a 5-point Likert scale at visit 2.
Safety and tolerability of Palomacare® vaginal gel | Through study completion, an average of 12 days
  To assess the safety and tolerability of Palomacare® vaginal gel using a 5-point Likert-type scale at visit 2 and by describing the incidence, nature and severity of adverse events (AEs) throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Santiago Palacios Gil-Antuñano, MD, Principal Investigator — Instituto Palacios de Salud y Medicina de la Mujer; Dr. Fernando Losa Domínguez, MD, Principal Investigator — Clínica Sagrada Familia
Locations (2):
- Spain (2):
  - Clínica Sagrada Familia, Barcelona
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid

IPD SHARING:
Plan to Share IPD: No
To be discussed